CLINICAL TRIAL: NCT04557410
Title: Open Label Study: Treatment of ALS Fatigue With PolyMVA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Band of Hope Foundation (Unknown)
Responsible Party: Principal Investigator, Raghav Govindarajan, Professor and Principal Investigator, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022342
Record Dates: First submitted 2020-05-31; First posted 2020-09-21 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving Supplement (Experimental): Participants receive supplement PolyMVA. Dose is 2 teaspoons twice a day.
  Interventions: Drug: PolyMVA

INTERVENTIONS:
Drug: PolyMVA — One-half teaspoon of PolyMVA contains the following:
  * Daily Value Thiamin (B-1) 23mg 1,533 Riboflavin (B-2) 0.45mg 26 Vitamin B-12 460mcg 7,666 Proprietary Blend 32mg - contains the following ingredients (no FDA value has been established on any of the following): Palladium, Alpha Lipoic Acid, Molybdenum, Rhodium, Ruthenium, Formyl Methionine, N-acetyl Cysteine.
  For each ml of Poly-MVA, the exact dosages are as follows:
  Palladium: 3.97mg Molybdenum: 0.044mg Ruthenium: 0.0014mg Rhodium: 0.014mg Lipoic Acid: 7.68mg Thiamine (B1): 9.26mg Riboflavin (B2): 0.174mg B12: 0.185mg Formyl Methionine: 0.026mg N-Acetyl cysteine: 0.185mg Vitamin A acetate 100 IU
  Other Ingredients: Distilled water, purified water, thiamine hydrochloride, Vitamin B12 as cyanocobalamin.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a disease that causes the death of upper and lower motor neurons. ALS symptoms are characterized by stiffness, muscle twitching, and worsening weakness due to muscle breakdown. Onset of symptoms are typically arm or leg weakness or difficulty speaking or swallowing and gradual development of overall body weakness. The cause is unknown and there is no cure for ALS.

Poly MVA was found to substantially lower fatigue and improve quality of life in a pilot study of patients with varied medical disorders. The reduction in fatigue was also observed in a small series of patients enrolled in an open label study for patients with gliomas.

In this study, we want to find out more about a dietary supplement, called Poly MVA (also called the study drug in this form), for people with ALS. We want to find out if Poly MVA reduces the symptoms of fatigue and depression when taken daily. The supplement contains vitamins, minerals and amino acids (proteins) and has been used by patients with other medical conditions to help with their fatigue and quality of life.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a disease that causes the death of upper and lower motor neurons. ALS symptoms are characterized by stiffness, muscle twitching, and worsening weakness due to muscle breakdown. Onset of symptoms are typically arm or leg weakness or difficulty speaking or swallowing and gradual development of overall body weakness. The cause is unknown and there is no cure for ALS.

Poly MVA is a dietary supplement which contains a uniquely formulated combination of minerals, vitamins, and amino acids designed to promote cellular energy production. The active molecule in this supplement is Palladium Lipoic Acid (PdLA) complex. This compound is synthesized using a process whereby palladium (a rare metal, which is found in the food chain- we consume approximately 2 ng/day is chemically bound to alpha lipoic acid, a powerful anti-oxidant involved in cellular energy.

Poly MVA was found to substantially lower fatigue and improve quality of life in a pilot study of patients with varied medical disorders. The reduction in fatigue was also observed in a small series of patients enrolled in an open label study for patients with gliomas.

Specific Aim 1: To test the efficacy of PolyMVA as a treatment for ALS fatigue.

Specific Aim 2: To determine the specificity of the fatigue reducing effect of Poly-MVA by controlling for mood, disease severity, and cognitive status

This is an open-label, prospective study which evaluates the response of 4 teaspoons of Poly MVA taken daily, over a 24-Week interval.

ELIGIBILITY:
Inclusion Criteria:

* Definite ALS
* Severe fatigue (defined by FSS > 4.0)
* Expanded Disability Status Scale (EDSS) (measure of neurological impairment) 0 - 7.5 Able to comply with study procedures
* Stable medication for the past month prior to enrollment.

Exclusion Criteria:

* na

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Change in fatigue severity | Baseline, 4 weeks, 8 weeks, 16 weeks, 20 weeks, 24 weeks
  Subjects will be assessed for fatigue using the Amyotrophic Lateral Sclerosis Functional Rating Scale - Respiratory (ALSFRS-R), a 12-item scale with possible scores ranging from 0 - 48 where 0 = total dependence and 48 = normal function.

SECONDARY OUTCOMES:
Change in impact of fatigue | Baseline, 4 weeks, 8 weeks, 16 weeks, 20 weeks, 24 weeks
  Modified Fatigue Impact Scale (MFIS), a 21-item rating scale with total scores ranging from 0 - 64 where the highest score reflects a greater impact of fatigue on a person's daily activity. Cam also be broken down into subscales: physical, cognitive, and psychosocial impacts.
Change in severity of depression | Baseline, 4 weeks, 8 weeks, 16 weeks, 20 weeks, 24 weeks
  Montgomery and Asberg Depression Rating Scale (MADRS), a scoring system used by the investigator based on a 10-item clinical interview moving from broadly phrased questions about symptoms to more detailed ones which allow a precise rating of severity. The rating are either given based on defined scale steps (0, 2, 4, 6) or between them (1,3,5), where higher scores indicate more severe depression (possible score is 0 - 60).

CONTACTS AND LOCATIONS:
Overall Officials: Raghav Govindarajan, MD, Principal Investigator — University of Missouri School of Medicine
Locations (1):
- University of Missouri-Columbia School of Medicine, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided